CLINICAL TRIAL: NCT04694144
Title: Results of Telescoping Nail in. OI; A Case Series
Brief Title: Results of Telescoping Nail In OI; a Case Series
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nariman Abol Oyoun, MD, Principal Investigator, Assiut University
Other Study IDs: TIN in osteogenesis
Record Dates: First submitted 2020-12-13; First posted 2021-01-05 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Osteogenesis Imperfecta
MeSH Terms: conditions — Osteogenesis Imperfecta

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: telescoping intramedullary nail — All osteogenesis imperfecta patients with lower limb skeletal deformities corrected with multiple corrective osteotomies and insertion of two parts male and female segments of intramedullary telescoping nail
  Other Names: growing nail

SUMMARY:
Assess the postoperative functional outcomes after surgical correction of skeletal deformities of lower limbs in osteogenesis imperfecta patients as regard ambulation status, postoperative complications and reoperation rate.

DETAILED DESCRIPTION:
Osteogenesis imperfecta (OI) is a rare heterogeneous group of inherited disorders characterized by brittle bones, frequent fractures, and skeletal deformities that affect an individual's ability to walk. Based on Sillence classification, there are four types of OI; Type I (mild, non-deforming), Type II (perinatal lethal), Type III (severely deforming), and Type IV (moderately deforming). Recently 3 types added type V, VI and type VII.

Deformities of the long bones are common in patients with osteogenesis imperfecta particularly in the lower limbs Where they are also more severe. Multiple fractures can occur and the ability to walk may be compromised.

The goal of orthopaedic surgery implies the correction of long bone bowing, rotational malalignment, angular deformity and prevention or reduction of the fracture incidence .Surgical intervention in the form of multiple osteotomies, realignment and fixation by intramedullary rods can correct deformity of the long bones and provides internal support enhancing the potential for standing and assisted or independent walking Sofield and Millar, Page and Mead popularized the operation of multiple osteotomies and fixation by intramedullary rods. In 1963 the baily dubow nail was first introduced The telescopic rodding and nailing have been developed in order to obtain a long lasting osteosynthesis in a growing long bone, thus, reducing the need of replacement. The evolution of telescoping rods for the treatment of fractures and deformity in children with diminished bone Quality has resulted in an approved and commercially available new single entry telescopic rod system, the Fassier Duval Telescopic IM System (FD-rod).

In recent publications a high reoperation rate for proximal rod migration and a complication rate up to 40% because of rod migration, limited telescoping and joint protrusion was found.

We hope that our study will advance the proper surgical intervention for children with osteogenesis imperfecta for better functional outcomes

ELIGIBILITY:
Inclusion Criteria:

* Age from 3-11 years
* Severe lower limb deformity presented with or without fracture

Exclusion Criteria:

* Nondisplaced/incomplete fractures in minimally deformed bones
* Deformity angulation less than 20 degree

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: all Osteogenesis imperfecta patients admitted at assiut university pediatric and main hospitals with age range 3- 11 years old presented with lower limb skeletal deformities with or without fracture will be included in our study
Sampling Method: Non-Probability Sample
Enrollment: 22 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Ambulation status | All patients will be assessed clinically and radiologically for deformity 6 months after surgery.
  the mobility status of each child will be allocated to one of the scores of the Gillette Functional Assessment Questionnaire Ambulation Scale and Hoffer and Bollock score
Rod Complications | All patients will be assessed radiologically for evidence of rod complications within the first two years after surgery.
  Radiographic evidence of rod problems including migration, bending, breakage, disengagement, jamming (failure of expansion/telescoping)

SECONDARY OUTCOMES:
Bone consolidation | All patients will be assessed clinically and radiologically one month after surgery.
  patients will be assessed for the average time in weeks of consolidation at the osteotomy site(s)
Timing of weight-bearing | All patients will be assessed clinically within the first three months after surgery.
  The average time in weeks until full weight bearing
Refracture | All patients will be assessed clinically and radiologically for refracture within the first two years after surgery.
  The occurrence of a second fracture at the same long bone with the rod in place or in association with any rod complication

OTHER OUTCOMES:
Knee Range of Motion | All patients will be assessed clinically for knee range of motion 6 months after surgery.
  The range within which the knee on the operated side can move in degrees

CONTACTS AND LOCATIONS:
Overall Officials: Nariman Abol Oyoun, MD, Lecturer, Principal Investigator — Assiut University
Locations (1):
- Assiut University Hospital AUH, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No